CLINICAL TRIAL: NCT05457790
Title: Feasibility and Preliminary Efficacy of Acceptance and Commitment Therapy (ACT) for Sleep Disturbances in Adults With Sickle Cell Disease (SCD): A Pilot Randomized Controlled Trial
Brief Title: Feasibility and Preliminary Efficacy of Acceptance and Commitment Therapy (ACT) for Sleep Disturbances in Adults With Sickle Cell Disease (SCD)
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Study on hold pending consideration for amendment.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 10000423; 000423-C
Record Dates: First submitted 2022-07-12; First posted 2022-07-14 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11-18

CONDITIONS: Sickle Cell Disease; Sickle Cell Anemia; Insomnia; Sleeplessness; Transient Insomnia; Nonorganic Insomnia; Chronic Insomnia
Keywords: Insomnia; Pain; Nonpharmacological; Actigraph; Anemia; Sleeplessness
MeSH Terms: conditions — Anemia, Sickle Cell; Sleep Initiation and Maintenance Disorders; Pain; Anemia | interventions — Waiting Lists

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1/Immediate Intervention Group (Active Comparator): 1-week baseline data collection period followed by an 8-week ACT intervention period focusing on acceptance, cognition defusion (i.e., not letting thoughts about sleep control behavior), present moment awareness, perspective taking, values, and committed actions.
  Interventions: Behavioral: ACT Intervention
- 2/Waitlist Control Group (Active Comparator): 1-week baseline data collection period followed by 8 weeks of maintaining usual routine followed by an 8-week intervention focusing on acceptance, cognition defusion (i.e., not letting thoughts about sleep control behavior), present moment awareness, perspective taking, values, and committed actions.
  Interventions: Behavioral: Waitlist

INTERVENTIONS:
Behavioral: ACT Intervention — 1-week baseline data collection period followed by an 8-week ACT intervention period focusing on acceptance, cognition defusion (i.e., not letting thoughts about sleep control behavior), present moment awareness, perspective taking, values, and committed actions.
  Arms: 1/Immediate Intervention Group
Behavioral: Waitlist — 1-week baseline data collection period followed by 8 weeks of maintaining usual routine followed by an 8-week intervention focusing on acceptance, cognition defusion (i.e., not letting thoughts about sleep control behavior), present moment awareness, perspective taking, values, and committed actions.
  Arms: 2/Waitlist Control Group

SUMMARY:
Research Type: Clinical Trial

Background:

People with sickle cell disease (SCD) have many health challenges. Also, they often have trouble sleeping. Acceptance and commitment therapy (ACT) might help people with SCD to improve their sleep problems.

Objective:

To see how well ACT works in people with SCD and sleep problems and to find out how they feel about it.

Eligibility:

People between the ages of 18 and 55 with SCD and trouble sleeping.

Design:

The study is remote. Participants will not have to come to the NIH at all. They will need a device that has Bluetooth and can connect to the internet.

Some participants will be in the study for 12 weeks. Others will participate for 20 weeks.

Participants will video chat with an ACT coach once a week for 8 weeks. The coach will guide participants through mindfulness exercises and teach ACT ideas. Each session lasts about 45 minutes.

Participants will be loaned an actigraph, a device worn on the wrist like a watch that measures and records movement. They will download a free app to upload data from the actigraph for the researchers.

Participants will wear the actigraph on their nondominant wrist day and night for either 4 or 6 designated weeks. During these weeks, participants will complete a sleep diary each morning when they wake up. This takes about 2 minutes.

Participants will be sent other surveys to complete from home during the study. They will answer questions about their physical and emotional health. These take 20-25 minutes.

The last survey will be 4 weeks after participants finish the ACT treatment. They will answer questions about how helpful they thought ACT was and how easy or hard it was to wear the actigraph.

DETAILED DESCRIPTION:
Background:

* Individuals with sickle cell disease (SCD) are faced with numerous challenges associated with their condition including sleep disturbance.
* Actigraphy is a wearable data collection device using accelerometry to track real-time body movements and is able to document several important aspects of sleep.
* Acceptance and Commitment Therapy (ACT) has been found effective in improving several aspects of health and wellbeing in individuals with chronic illness and pain, including sleep disturbance.
* To our knowledge, ACT for sleep disturbance has not been investigated yet among individuals with SCD.

Objective:

To assess the feasibility and acceptability of an ACT for Sleep intervention in adults with SCD.

Eligibility:

* Adults (>=18 - <=55) with a self-reported diagnosis of sickle cell disease.
* Access to necessary resources for participating in a technology-based intervention (i.e., computer, tablet, or smartphone with internet access).
* Must score a T-score of 57.5 or higher from the PROMIS(R) (Patient-Reported Outcomes Measurement Information System(R) Sleep Disturbance Scale.
* Ability to read and speak English.

Design:

* This is a pilot randomized controlled trial (RCT) comparing participants who receive an 8-week ACT intervention (n = 15) with those in a wait-list control group (n = 15). We will aim to recruit three additional participants for each group to allow for dropouts, so our total target accrual is 36.
* The study requires a 1-week baseline actigraphy data collection period followed by an 8-week ACT intervention period.
* The intervention period includes four one-on-one approximately 60-minute sessions with a psychologist or psychology associate over an NIH-approved telehealth platform.
* Participants will wear an actigraphy monitor on non-dominant wrists during designated data collection periods. Participants also will complete measures on health and well-being (e.g., sleep, cognitive functioning, quality of life, and experiential avoidance) at preintervention, post-intervention, and a 1-month follow-up assessment.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Ability of participant to understand and the willingness to sign a written informed consent document
* Ability to read and speak English
* Age >=18 - <= 55 years
* Self-reported active diagnosis of Sickle Cell Disease
* Must score a T-score of 57.5 or higher from the PROMIS Sleep Disturbance Scale
* Self-reported sleep disturbance of at least 3 months
* Access to necessary resources for participating in a technology-based intervention (i.e., computer, smartphone or tablet with internet access and either a USB port or Bluetooth capability)
* Must be willing to register online and install the software to use the actigraph and willing to complete the sleep diaries
* Must be able and willing to attend remote ACT coaching calls during the study team s working hours

EXCLUSION CRITERIA:

* Uncontrolled psychiatric illness, cognitive impairments, or other circumstance as judged by the Principal Investigator (PI) or Lead Associate Investigator (LAI), both licensed psychologists, that would limit compliance with study requirements
* Evidence of disease progression at the time of referral to this study to the extent that it would impede participation or completion of evaluations as determined by the medical advisory investigator in conjunction with the study PI/LAI
* Individuals who are planning to start a new treatment or who are planning to change medications (e.g., pharmacological, dietary supplements, or psychological) for sleep disturbance or that have been known to significantly affect sleep in the next 6 months (Current sleep medication is not an exclusion criteria)
* Individuals currently enrolled in a treatment protocol that would impact sleep
* Previous treatment that cured sickle cell disease.
* Individuals scheduled to receive gene therapy or stem cell therapy, or begin the conditioning regimen for these procedures, in the next 6 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2024-05-03 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility | Weeks 4, 8, and 12
  (i) Treatment specific retention rate among all randomized participants, with a target retention rate of 70% over the 8-week intervention period (excluding those who are taken off study due to extended/frequent hospitalizations or disease complications). (ii) Compliance with at-home ACT practices per sleep diary, with a target of 4 days per week on average as assessed by a daily question during weeks 4, 8, and 12.
Acceptability | 4 Weeks post intervention
  Patient responses on the Acceptability questionnaire; a mean score >3.0 on items 1-4 will be deemed to reflect adequate satisfaction.

SECONDARY OUTCOMES:
Relationships among sleep, pain, and quality of life at baseline. | Baseline
  We will assess correlations between sleep variables (as described above), pain (PROMIS-57 pain scales), and the remaining PROMIS-57 quality of life subscales.
Relationship between objective and subjective measures of sleep in SCD. | Baseline, Weeks 4, 8, and 12
  We will assess the correlations between sleep variables obtained with diaries and actigraphy (i.e., total sleep time, sleep efficiency, sleep onset latency, and wake after sleep onset).

CONTACTS AND LOCATIONS:
Overall Officials: Staci M Peron, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000423-C.html